CLINICAL TRIAL: NCT05781958
Title: Cadonilimab Combined With Gemcitabine and Cisplatin as First Line Therapy in Patients With Advanced Intrahepatic Cholangiocarcinoma: A Single Center, Single Arm, Phase II Trial
Brief Title: Cadonilimab Combined With Gem/Cis as First Line Therapy in Patients With Advanced ICC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shen Feng (Other)
Responsible Party: Sponsor-Investigator, Shen Feng, Professor and Chief Surgeon, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBHKY2022-H039-P001
Record Dates: First submitted 2023-02-20; First posted 2023-03-23 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: cadonilimab (anti-PD-1/CTLA-4 bispecific antibody)
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+Gem/Cis (Experimental)
  Interventions: Drug: Cadonilimab+Gem/Cis

INTERVENTIONS:
Drug: Cadonilimab+Gem/Cis — Cadonilimab (500mg, iv, Q3W, Day1) with gemcitabine(1000mg/m^2, iv, Q3W, Day1and Day8) plus cisplatin(25mg/m^2, iv, Q3W, Day1and Day8) up to 8 cycles followed by cadonilimab (500mg, iv, Q3W, Day1) plus capecitabine（1000 mg/m^2 orally according to Body Surface Area (BSA)，BID，Q3W，on Days 1-14）as maintenance therapy until disease progression or other discontinuation criteria, up to 24months.

SUMMARY:
TOPAZ-1 phase III trail demonstrated that the addition of immune checkpoint inhibitor anti-PD-L1 antibody improved progression-free survival (PFS) and overall survival (OS) compared to Gem/Cis alone. Cadonilimab is a first-in-class bispecific, humanized IgG1 antibody targeting PD-1 and CTLA-4, which has the potential to boost immune surveillance in tumors. The goal of this clinical trial is to evaluated the efficacy and safety of cadonilimab combined with gemcitabine and cisplatin as first Line therapy in patients with advanced intrahepatic cholangiocarcinoma. Eligible participants will receive cadonilimab (up to 12 months) plus gemcitabine and cisplatin (for maximum of 6-8 cycles) until radiologic disease progression, unacceptable toxicity, or withdrawal from the study, whichever occurred first. The primary endpoint is objective response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed intrahepatic cholangiocarcinoma (ICC)
2. At least 1 measurable lesion (according to RECIST1.1)
3. Have not previously received any systemic treatment
4. Age 18-75 years old, both male and female
5. ECOG performance status score (PS score) 0-2 point
6. Adequate medullary hematopoiesis function: Neutrophils≥1.5*10^9/L; platelets≥100*10^9/L
7. Adequate renal function: creatinine clearance > 60ml/min
8. Adequate hepatic function: Bilirubin ≤ 1.5 times the upper limit of normal
9. No cardiac insufficiency or chest pain (medically uncontrollable); no myocardial infarction in the 12 months prior to study initiation
10. Expectation survival time over 3 months
11. The patient must sign an informed consent form

Exclusion Criteria:

1. History of another primary malignancy
2. Brain metastases or spinal cord compression
3. Uncontrolled intercurrent illness
4. Have active or previously recorded autoimmune or inflammatory diseases (eg Rheumatoid arthritis, psoriasis, systemic lupus erythematosus, AIDS, etc)
5. Have received allogeneic organ transplantation
6. Control of concurrent complications, including but not limited to persistent or active infections, symptomatic congestive heart failure, poorly controlled hypertension, unstable angina, poorly controlled arrhythmia, active interstitial lung disease ( ILD), severe chronic gastrointestinal disorders associated with diarrhea symptoms, may limit compliance with the psychiatric/social conditions required by the trial, and substantially increase the risk of adverse events or affect the ability of patients to sign written consent forms
7. History of active primary immunodeficiency
8. Pregnant or lactating women
9. Severe or uncontrolled infections
10. Patients with history of severe neurological or psychiatric illness, including dementia or epilepsy;
11. Patients with drug abuse, medical, psychological or social conditions that may interfere with the study results or the assessment of the study results;
12. Patients are unsuitable for the enrollment according to investigator's judgement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per RECIST 1.1 | Up to two years
  Defined as patients achieving a complete response [CR] or partial response [PR]

SECONDARY OUTCOMES:
Progression free survival (PFS) per RECIST 1.1 | Up to two years
  Defined as the time from the start of treatment to the date of progressive disease, or death, whichever occurred first.
Desease control rate (DCR) per RECIST 1.1 | Up to two years
  CR + PR + SD
Overall survival (OS) | Up to two years
  Defined as the time from the start of treatment to the date of death from any cause
6mo PFS rate per RECIST 1.1 | at 6 months
  Progression-free survival (PFS) rate at 6 months
adverse events | Up to two years
  Include Treatment emerge adverse events, treatment related adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China